CLINICAL TRIAL: NCT02872623
Title: EnteroCT With Enteroclysis Versus Enterography-MRI for the Diagnosis of Tumors of the Small Intestine: a Pilot Study
Acronym: enteroMRI-TSI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PO14065
Record Dates: First submitted 2016-08-16; First posted 2016-08-19 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Suspicion of Tumor of the Small Intestine

ARMS (1):
- experimental group (Experimental): patients clinically suspected of having a tumor of the small intestine
  Interventions: Radiation: Enterography-MRI without enteroclysis; Radiation: enteroCT with enteroclysis

INTERVENTIONS:
Radiation: Enterography-MRI without enteroclysis
Radiation: enteroCT with enteroclysis

SUMMARY:
Early diagnosis of tumors of the small intestine is a challenge for clinicians and for radiologists. The detection of tumors of the small intestine is a field in which the video capsule endoscopy has the lowest performance.

The entero-CT with enteroclysis is the imaging technique used primarily to explore patients with a strong suspicion of small intestine tumors. However the entero-CT with enteroclysis has disadvantages : it is irradiating, the nasojejunal tube implies a discomfort to the patient and it is a complicated examination in terms of logistics with necessity of specific equipment to insert the nasojejunal tube.

MRI has been proposed as an alternative imaging technique and satisfactory results have been reported with the MRI enteroclysis. However, this technique has several disadvantages related to nasojejunal tube insertion and the necessity of equipment compatible with the high magnetic fields. The enterography-MRI without enteroclysis, whose principle is to distend the small intestine by ingestion of large quantities of a liquid, has a major and undisputed role in the exploration of Crohn's disease of the small bowel. However, its capacity for distension of the small intestine for optimal tumor detection is questioned and its role in tumor detection is largely unknown.

DETAILED DESCRIPTION:
Evaluate the diagnostic performances of enteroCT with enteroclysis and enterography-MRI without enteroclysis, for the diagnosis of tumor of the small intestine, among patients with suspicion of small intestine tumors.

ELIGIBILITY:
Inclusion Criteria:

* patient clinically suspected of having a tumor of the small intestine
* patient consenting to participate to the study
* patient enrolled in the national healthcare insurance program
* patient older than 18 years

Exclusion Criteria:

* patient with inflammatory bowel disease
* patient with contraindication for MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-03; Primary Completion 2018-03 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Presence of a tumor of the small intestine | 12 months
  Presence of a tumor of the small intestine diagnosed using pathological results or using clinical evaluation at 12 months (if no biopsy is performed).

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Reims, Reims, France, France